CLINICAL TRIAL: NCT06260813
Title: Biomechanical and Morphological Characterization of the Foot in Patients With Posterior Tibial Tendon Dysfunction.
Brief Title: Biomechanical and Morphological Characterization of PTTD
Acronym: PTTD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S66277
Record Dates: First submitted 2023-12-08; First posted 2024-02-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Posterior Tibial Tendon Dysfunction
MeSH Terms: conditions — Posterior Tibial Tendon Dysfunction | interventions — Radiography; Ultrasonography; Tomography, X-Ray Computed; Gait Analysis

STUDY DESIGN:
Intervention Model Description: Prospective interventional study that includes PTTD patients (PTTD I, II and III) and a healthy control group.
Who Masked: Participant
Masking Description: PTTD patients (PTTD I, II and III) and a healthy control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTTD patients (PTTD I, II and III) (Experimental): 75 patients with PTTD (25 patients in Stage I, 25 patients in Stage II, 25 patients in Stage III)
  Interventions: Diagnostic Test: Radiography; Diagnostic Test: Ultrasound; Diagnostic Test: MRI; Diagnostic Test: CT-scan; Diagnostic Test: Gait analysis
- Healthy control group (Experimental): 25 healthy volunteers
  Interventions: Diagnostic Test: Radiography; Diagnostic Test: CT-scan; Diagnostic Test: Gait analysis

INTERVENTIONS:
Diagnostic Test: Radiography — X-rays of the ankle; anterior-posterior, lateral, Mortise view and hindfoot alignment view. Standard weight bearing x-rays of the foot; anterior-posterior, lateral and oblique view.
Diagnostic Test: Ultrasound — Ultrasound of the posterior tibial tendon to see if there is an irritation, elongation or rupture.
  Arms: PTTD patients (PTTD I, II and III)
Diagnostic Test: MRI — MRI when ultrasound is not conclusive to identify an irritation, elongation or rupture of the posterior tibial tendon.
  Arms: PTTD patients (PTTD I, II and III)
Diagnostic Test: CT-scan — CT-scan to identify arthritis of the tibial-talar, subtalar and/or Chopart joints.
Diagnostic Test: Gait analysis — This lab is equipped with a 10-meter walkway surrounded by a passive optoelectronic motion analysis system consisting of 10 cameras to track the motion of markers. In the middle of the walkway, a force plate is integrated, with a pressure plate placed on top.

SUMMARY:
Posterior tibial tendon dysfunction (PTTD) is a progressive condition of the tendon of the tibialis posterior muscle with symptoms of tendinopathy or even rupture. Functionally, it is associated with the inability to lock the mid foot and thus manifests itself as a main contributor to adult acquired flatfoot deformity.

Concerning treatment, clinical decision making is currently based on a classification integrating various parameters as pain, flexibility of the foot joints, the condition of the posterior tibial tendon assessed through ultrasound imaging and radiographic assessment of arthritic changes. Surprisingly, this classification does not consider any morphologic characteristics (the shape of a bone or joint) or functional, biomechanical characteristics of the foot and ankle, i.e. based on kinematics (e.g. range of motion) and/or kinetics (center of pressure, angular velocity, moment, power absorption and power generation of a joint).

Detailed biomechanical characteristics of the foot and ankle can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform. Kinematic studies in the field of PTTD typically considered the foot as a structure consisting of three segments: hind foot, forefoot and hallux. Consequently, the mid foot segment (the Chopart and Lisfranc joints) has been neglected, although it is this segment that is particularly affected in PTTD patients.

The aim of this research is to overcome the limitations of the current classification system and treatment of PTTD patients, by complementing the current standard-of-care clinical assessment with better insight in the pathologic changes that occur in PTTD patients.

DETAILED DESCRIPTION:
Posterior tibial tendon dysfunction (PTTD) is a progressive condition of the tendon of the tibialis posterior muscle with symptoms of tendinopathy or even rupture. Functionally, it is associated with the inability to lock the mid foot and thus manifests itself as a main contributor to adult acquired flatfoot deformity. Importantly, this condition is associated with severe pain, inability to walk, collapse of the foot arch and dislocation and destruction of foot joints, causing serious disability with respect to activities of daily living and professional activities.

Concerning treatment, clinical decision making is currently based on a classification integrating various parameters as pain, flexibility of the foot joints, the condition of the posterior tibial tendon assessed through ultrasound imaging and radiographic assessment of arthritic changes. PTTD stage 1 is characterized by tendinopathy and is suggested to be mainly treated conservatively. Stage 2 is characterized by a flexible flat foot deformation, mostly combined with a tear of the posterior tibial tendon. Here, treatment is suggested through osteotomies and soft tissue surgery. Stage 3 encompasses a rigid flat foot deformity associated with a fully dysfunctional posterior tibial tendon and degenerative changes of the hind foot joints. At this stage fusion of the affected joints should be considered. During recent decades, this classification has been extended with additional subgroups as well as a stage 4 which adds onto stage 3 with excessive tibio-talar valgus and is mainly treated by a complementary fusion of the ankle joint.

Surprisingly, this classification does not consider any morphologic characteristics (the shape of a bone or joint) or functional, biomechanical characteristics of the foot and ankle, i.e. based on kinematics (e.g. range of motion) and/or kinetics (center of pressure, angular velocity, moment, power absorption and power generation of a joint).

Detailed biomechanical characteristics of the foot and ankle can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform. Kinematic studies in the field of PTTD typically considered the foot as a structure consisting of three segments: hind foot, forefoot and hallux. Consequently, the mid foot segment (the Chopart and Lisfranc joints) has been neglected, although it is this segment that is particularly affected in PTTD patients. While kinematic studies focus on joint motion, kinetic studies focus on the loading and impact associated with motion of the joints.

Besides documenting specific biomechanical characteristics of the different stages of PTTD, it is essential to explore the relation of these biomechanical characteristics with the bone morphology of the involved osseous structures.

The aim of this research is to overcome the limitations of the current classification system and treatment of PTTD patients, by complementing the current standard-of-care clinical assessment with better insight in the pathologic changes that occur in PTTD patients. This will be done by simultaneously acquiring kinematic, kinetic and morphologic characteristics in PTTD patients, with a special interest in the possible connection between these morphological and the biomechanics changes. Through these insights, we will be able to better classify these patients, using the developed biomechanical classification, as a first step towards an optimized, patient-tailored treatment plan which converts these individual pathological characteristics back to normal, giving the patients back their mobility and a live without pain, i.e. gaining back their quality of life.

ELIGIBILITY:
Inclusion criteria:

* Patient groups:

  * Posterior tibial tendon dysfunction (all clinical stages)
  * Age 18-675 year
  * ICF obtained
* Control group:

  * No pain complaints
  * No pes plano valgus, PTTD or pes cavo varus or other foot and ankle pathology
  * Age 18-75 year
  * ICF obtained

Exclusion criteria patient and control groups:

* Being younger than 18 years
* Inability to walk without mobility aids
* Inability to walk < 100 meter
* Difference in leg length > 3cm
* Subjects with BMI>30 kg/m², due to less accurate gait analysis by absence of anatomical landmarks
* Subjects unable to perform a gait analysis
* Any medical condition possibly affecting normal gait.
* Pregnancy: at the start or during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Kinematic characteristics during Gait analysis | 1 year
  Range of Motion (ROM) of PTTD patient of each stage will be obtained and compared between the patient groups (PTTD 1-2-3) and a control group.
Center of pressure during Gait analysis | 1 year
  The center of pressure (kinetic characteristic) of PTTD patients of each stage will be obtained and compared between the patient groups (PTTD 1-2-3) and a control group. This information can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform.
Angular velocity during Gait analysis | 1 year
  The angular velocity (kinetic characteristic) of PTTD patients of each stage will be obtained and compared between the patient groups (PTTD 1-2-3) and a control group. This information can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform.
Moment during Gait analysis | 1 year
  The moment (kinetic characteristic) of PTTD patients of each stage will be obtained and compared between the patient groups (PTTD 1-2-3) and a control group. This information can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform.
Power absorption during Gait analysis | 1 year
  The power absorption (kinetic characteristic) of PTTD patients of each stage will be obtained and compared between the patient groups (PTTD 1-2-3) and a control group. This information can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform.
Power generation during Gait analysis | 1 year
  The power generation (kinetic characteristic) of PTTD patients of each stage will be obtained and compared between the patient groups (PTTD 1-2-3) and a control group. This information can be reliably collected by instrumented gait analysis wherein a 3D camera system is combined with a force plate and plantar pressure platform.
Bone morphology | 1 year
  Morphological characteristics of PTTD patients of each stage will be obtained by CT-scan and statistical shape modeling and compared between the study groups and a control group.

SECONDARY OUTCOMES:
American Orthopaedic Foot & Ankle Society (AOFAS) score | 1 year
  Patients Reported Outcome Measures. It combines five patient-reported items concerning pain and function with four physician-determined items concerning function and alignment, on a 0 to 100-point scale with healthy ankles receiving 100 points.
European Foot and Ankle Society (EFAS) score | 1 year
  Patients Reported Outcome Measures consisting of six questions on pain and function. A total of 24 points can be achieved on a 5-point scale (0-4), whereby a high score means a good result.
36-item Short Form Health Survey (SF36) | 1 year
  Patients Reported Outcome Measures that measures health-related quality of life and health care needs. The instrument includes scales for physical functioning, social functioning, role limitations due to physical or emotional problems, mental health, energy, pain and general health perception. A high score corresponds to better health status.
Visual Analogue Scale (VAS) pain | 1 year
  Patients Reported Outcome Measures to quantify the pain of a patient. The VAS pain score runs from 10 to 0, where 10 is "Worst possible pain" and 0 is "No pain".
Visual Analogue Scale (VAS) satisfaction | 1 year
  Patients Reported Outcome Measures to quantify the satisfaction of a patient. The VAS satisfaction score runs from 10 to 0, where 10 is "Very satisfied" and 0 is "unsatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Sander Wuite, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No